CLINICAL TRIAL: NCT00981773
Title: A Prospective, Randomised Study to Assess Safety, Changes in Platelet Reactivity, Plasma Cardiac Biomarkers, Immunological and Metabolic Parameters in HIV-1 Infected Subjects Undergoing a Switch in Antiretroviral Therapy
Brief Title: The St. Marys and The Mater Switch Study
Acronym: SMASH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment problem
Sponsor: Imperial College London (Other)
Collaborators: Mater Misericordiae University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0 18.6.2009
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections
Keywords: HIV switch; HIV; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate switch (Experimental): * Continue current boosted protease inhibitor
  * Switch NRTI backbone to maraviroc 150 mg bid
  Interventions: Drug: Maraviroc
- Continue current antiretroviral therapy (Active Comparator): * Continue current antiretroviral regimen until week 12 then switch therapy as per arm 1.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 150 mg bid
  Arms: Immediate switch
Drug: Maraviroc — maraviroc 150 mg bid switch 12 weeks later
  Arms: Continue current antiretroviral therapy

SUMMARY:
The aim of the study is to determine whether switching from an antiretroviral regimen containing abacavir and/or didanosine to one containing maraviroc will lead to a reduction in platelet reactivity and inflammatory markers at weeks 12 and 24 thereby conferring a reduction in cardiac risk.

In addition the study will assess the efficacy of a maraviroc containing regimen in combination with a boosted protease inhibitor in terms of tolerability and achieving long term viral suppression as assessed at week 48.

The investigators hypothesize that there will be a rapid reduction in platelet reactivity on switching to maraviroc and that a boosted protease inhibitor in combination with maraviroc will provide a safe and efficacious antiretroviral regimen enabling a reduction in cardiac risk whilst maintaining virological suppression.

DETAILED DESCRIPTION:
To assess the safety, changes in platelet reactivity, plasma cardiac biomarkers and metabolic parameters in HIV 1 infected subjects undergoing a switch in ART from a nucleoside containing regimen which includes abacavir and / or didanosine to a maraviroc containing regimen.

40 HIV-1 infected subjects currently receiving stable antiretroviral therapy consisting of a boosted protease inhibitor and two NRTIs including abacavir and / or didanosine will be recruited. Subjects will be randomized on a 1:1 basis to one of two arms:

Arm 1 (immediate switch in antiretroviral therapy)

* Continue current boosted protease inhibitor
* Switch NRTI backbone to maraviroc 150 mg bid

Arm 2 (continue current antiretroviral therapy)

* No change to current antiretroviral therapy for twelve weeks
* After twelve weeks switch therapy as per Arm 1

Subjects will be followed up for 48 weeks and will attend for clinic visits at screening, baseline, weeks 4, 12, 16, 24, 36 and 48. Platelet reactivity, inflammatory and cardiac biomarkers and markers of T cell activation will be assessed at baseline, week 12 and week 24.

Following completion of the study subjects may continue their study antiretroviral regimen or switch to an alternative regimen at their clinician's discretion.

Inclusion Criteria

* HIV-1 infected males or females
* Between 18 and 65 years of age
* Signed informed consent
* Currently receiving a stable antiretroviral regimen comprising of:

  * two licensed NRTIs including abacavir and/or didanosine
  * any licensed boosted protease inhibitor at any dose (excluding tipranavir*)
* Undetectable plasma HIV RNA to less than 50 copies/mL for at least 24 weeks prior to screening
* Availability of stored plasma with which to perform a tropism assay
* CCR5 tropic HIV virus based on a tropism assay from a stored plasma sample
* Willing to continue unchanged, or to modify antiretroviral therapy, in accordance with the randomisation assignment
* No documented viral resistance to currently licensed HIV-1 protease inhibitors based either on previous HIV-1 genotypic resistance testing or in the judgement of the study investigators
* No previous exposure to maraviroc or CCR5 receptor antagonists
* Subjects in good health upon medical history, physical exam, and laboratory testing in the opinion of the investigator
* Female subjects who are heterosexually active and of childbearing potential (i.e., not surgically sterile or at least two years post menopausal) must avoid becoming pregnancy as follows from screening through completion of the study using one or both of the following methods:

  * barrier contraceptives (condom, diaphragm with spermicide)
  * IUD PLUS a barrier contraceptive
* Female subjects of childbearing potential must have a negative pregnancy test. Exclusion criteria
* failure of current antiretroviral regimen due to virological failure
* active opportunistic infection, malignancy or significant co-morbidities in the opinion of the investigator
* pregnancy
* current prohibited concomitant medication (as listed in section 4.1.4)
* no available stored plasma sample predating their current antiretroviral regimen upon which a tropism assay can be performed
* active HBV infection as evidenced by positive hepatitis B surface antigen
* active hepatitis C virus infection as evidenced by positive HCV PCR or HCV antibody

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected males or females
* Between 18 and 65 years of age
* Signed informed consent
* Currently receiving a stable antiretroviral regimen comprising of:

  * two licensed NRTIs including abacavir and/or didanosine
  * any licensed boosted protease inhibitor at any dose (excluding tipranavir*)
* Undetectable plasma HIV RNA to less than 50 copies/mL for at least 24 weeks prior to screening
* Availability of stored plasma with which to perform a tropism assay
* CCR5 tropic HIV virus based on a tropism assay from a stored plasma sample
* Willing to continue unchanged, or to modify antiretroviral therapy, in accordance with the randomisation assignment
* No documented viral resistance to currently licensed HIV-1 protease inhibitors based either on previous HIV-1 genotypic resistance testing or in the judgement of the study investigators
* No previous exposure to maraviroc or CCR5 receptor antagonists
* Subjects in good health upon medical history, physical exam, and laboratory testing in the opinion of the investigator
* Female subjects who are heterosexually active and of childbearing potential (i.e., not surgically sterile or at least two years post menopausal) must avoid becoming pregnancy as follows from screening through completion of the study using one or both of the following methods:

  * barrier contraceptives (condom, diaphragm with spermicide)
  * IUD PLUS a barrier contraceptive
* Female subjects of childbearing potential must have a negative pregnancy test

Exclusion Criteria:

* failure of current antiretroviral regimen due to virological failure
* active opportunistic infection, malignancy or significant co-morbidities in the opinion of the investigator
* pregnancy
* current prohibited concomitant medication (as listed in section 4.1.4)
* no available stored plasma sample predating their current antiretroviral regimen upon which a tropism assay can be performed
* active HBV infection as evidenced by positive hepatitis B surface antigen
* active hepatitis C virus infection as evidenced by positive HCV PCR or HCV antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in platelet reactivity between treatment arms at week 12 | 48 weeks

SECONDARY OUTCOMES:
To assess for the following: Mean change over 24 weeks and mean difference at week 12 between study groups in plasma inflammatory and cardiac biomarkers and markers of immune activation | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, MBChB, Principal Investigator — Imperial College London; Patrick Mallon, MBChB, Principal Investigator — UCD School of Medicine and Medical Sciences
Locations (3):
- Ireland (2):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
- Imperial College Healthcare NHS Trust, London, United Kingdom